CLINICAL TRIAL: NCT02678871
Title: Combined Transcatheter Aortic Valve Implantation and Percutaneous Closure of the Left Atrial Appendage
Acronym: TAVI-LAAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device was withdrawn from the market
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01-18
Record Dates: First submitted 2016-01-28; First posted 2016-02-10 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Aortic Valve Disorder
Keywords: Aortic Valve Stenosis; Left atrial appendage
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All study participants (Other): Patients meeting clinical and anatomical pre-requisites will undergo TAVI with the LOTUS or Acurate Neo heart valve system (or subsequent CE marked iterations) and LAA closure with the WATCHMAN device in the same setting. Dual antiplatelet therapy (clopidogrel and acetylsalicylic acid) will be prescribed for 6 months followed acetylsalicylic acid indefinitely. Follow-up will be performed after 1 month, 6 months and 1 year.
  Interventions: Device: Lotus or ACURATE neo Heart valve system (or subsequent CE marked iterations); Device: WATCHMAN

INTERVENTIONS:
Device: Lotus or ACURATE neo Heart valve system (or subsequent CE marked iterations) — Patients meeting clinical and anatomical pre-requisites will undergo TAVI with the Lotus or ACURATE neo Heart valve system (or subsequent CE marked iterations)
Device: WATCHMAN — LAA closure with the WATCHMAN device

SUMMARY:
Atrial fibrillation (AF) is a common comorbidity of patients candidates to transcatheter aortic valve implantation (TAVI). The management of chronic oral anticoagulation (OAC) for the prevention of ischemic stroke is very challenging in this population of complex and frail subjects. Since the percutaneous left atrial appendage (LAA) closure with the WATCHMAN device proved promising safety and efficacy results in randomized comparisons with OAC (current standard of care), the aim of the current study is to assess the feasibility and the early safety of performing TAVI with the Lotus System and percutaneous LAA closure with the WATCHMAN device at the same session.

ELIGIBILITY:
Inclusion Criteria:

* TAVI candidates
* Elderly patients with symptomatic, severe, calcific, native aortic valve stenosis, assessed by echocardiography AVA up to 1.0 cm2 or AVAi up to 0.6 cm2m2 and mean pressure gradient 40 mmHg or jet velocity 4 ms
* Inoperable or at increased surgical risk (according to multidisciplinary heart team decision)
* Non-valvular AF (paroxysmal, persistent or permanent)
* CHA2DS2-VASc ≥ score
* HAS-BLED score ≥ 2
* Written informed consent
* Aortic annulus size ≥ 20 mm and ≤ 27 mm
* Adequate LAA ostium diameter (17 31mm)

Exclusion Criteria:

* Previous TAVI
* Previous LAA closure (surgical or percutaneous)
* Previous RF ablation of AF
* Need for long-term OAC (history of pulmonary embolism, mechanical heart valve)
* Contraindication to aspirin
* Relevant CAD requiring revascularization
* Infective endocarditis
* LV ejection fraction < 20 percent
* Cardiogenic shock or hemodynamic instability
* Symptomatic carotid disease
* Life expectancy < 1 year
* Severe renal failure (dialysis or serum creatinine level > 3.0 mg/dl or 265 μmol/L)
* CVE within the past 3 months
* Acute complications occurring during TAVI procedure
* Congenital unicuspid aortic valve
* Femoral artery lumen diameter <6.0 mm or <6.5 mm (for the 23-mm valve or the 25-mm and 27-mm valves, respectively)
* Documented LAA and/or LV thrombi
* Severe MR
* Atrial septal defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Early safety (composite endpoint of TAVI-related (according to VARC 2 criteria) and percutaneous LAA closure-related events at 30 days) | 30 Days
  Early safety - composite endpoint of TAVI-related (according to VARC 2 criteria) and percutaneous LAA closure-related events at 30 days. Composite defined as all cause-mortality, all stroke (disabling and non-disabling), life threatening bleeding, acute kidney injury (stage 2 or 3, including renal replacement therapy), coronary artery obstruction requiring intervention, major vascular complications, valve-related dysfunction requiring repeat procedure, pericardial effusion requiring pericardial drainage, and LAA device embolization requiring surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, Prof. Dr., Principal Investigator — Inselspital Bern, Universitätsklinik für Kardiolgie
Locations (6):
- Universitätsmedizin Rostock Zentrum für Innere Medizin Abteilung für Kardiologie, Rostock, Germany
- Italy (3):
  - Structural Heart Disease Interventions Unit - IRCCS Policlinico San Donato, San Donato Milanese, Milano
  - Azienda Ospedaliera Universitaria Policlinico "G.Rodolico ", Catania
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Santa Maria University Hospital,, Lisbon, Portugal
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No